CLINICAL TRIAL: NCT07220200
Title: A Prospective, Multi-Site, Interventional Case-Series Evaluating the MOVE (Movement-Oriented Velocity of Engagement) Protocol for Musculoskeletal Pain Recovery
Brief Title: MOVE Protocol - Movement-Oriented Velocity of Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MMSx Authority Institute for Movement Mechanics and Biomechanics Research Inc (Unknown)
Responsible Party: Sponsor
Organization: MMSx Authority Institute for Movement Mechanics & Biomechanics Research Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOVE-001/2025
Record Dates: First submitted 2025-10-22; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Musculoskeletal Pain - Acute and Subacute Conditions
Keywords: Rehabilitation Biomechanics Early Mobilization Movement Therapy Functional Recovery Pain Management Physical Therapy

STUDY DESIGN:
Intervention Model Description: This was a multi-site, single-arm interventional case-series evaluating the MOVE (Movement-Oriented Velocity of Engagement) rehabilitation protocol for acute and subacute musculoskeletal pain. Forty participants across four international centers completed an 8-week standardized intervention consisting of four progressive phases: Mobilize, Optimize Load, Validate Neural Control, and Energize Recovery. The study aimed to assess safety, functional recovery, and pain reduction outcomes following the MOVE protocol.
Masking Description: Open-label rehabilitation study. Both investigators and participants were aware of the intervention procedures, as exercise-based protocols require therapist supervision and participant engagement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Move Protocol (Experimental): Participants received the MOVE (Movement-Oriented Velocity of Engagement) rehabilitation protocol, consisting of four progressive phases: Mobilize, Optimize Load, Validate Neural Control, and Energize Recovery. The program emphasized functional movement restoration, load tolerance, and neuromuscular coordination.
  Interventions: Behavioral: MOVE Rehabilitation Protocol

INTERVENTIONS:
Behavioral: MOVE Rehabilitation Protocol — The MOVE (Movement-Oriented Velocity of Engagement) protocol is a biomechanics-based rehabilitation approach targeting early mobilization and functional recovery for musculoskeletal pain conditions. The structured program includes four key phases: Mobilize, Optimize Load, Validate Neural Control, and Energize Recovery, applied over 8 weeks under therapist supervision.

SUMMARY:
A Prospective, Multi-Site, Interventional Case-Series Evaluating the MOVE (Movement-Oriented Velocity of Engagement) Protocol for Musculoskeletal Pain Recovery

DETAILED DESCRIPTION:
The MOVE Protocol is a structured, biomechanics-based rehabilitation framework designed to accelerate recovery from musculoskeletal pain conditions through progressive mobilization and neuromuscular control. This interventional case-series involved multiple clinical and training centers (BodyGNTX, GFFI, IIKBS, ASFU) and applied standardized MOVE sessions under the supervision of certified movement specialists. Assessments included pain scoring (NRS), functional mobility (LEFS/UEFI), and balance control, measured at baseline, week 2, week 4, and week 8. The protocol followed ICH-GCP E6(R2) and Helsinki 2013 guidelines, with institutional ethics approval from MMSx Authority IREB. The study demonstrated safe and effective early-movement outcomes across diverse populations, emphasizing mobility, load optimization, and neuromuscular revalidation.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18-65 years diagnosed with acute or subacute musculoskeletal pain or movement restriction (≤12 weeks duration).

  * Capable of performing supervised rehabilitation and daily movement tasks.
  * Able to provide informed consent and comply with study assessments.
  * Baseline pain score ≥4 on the Numerical Rating Scale (NRS).

Exclusion Criteria:

* Chronic pain (>12 weeks) or neurological disorders affecting movement control.

  * Post-surgical cases or fractures within the past 3 months.
  * Cardiopulmonary or systemic illness contraindicating exercise participation.
  * Pregnancy or conditions limiting safe participation in physical rehabilitation.
  * Refusal to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Pain Reduction (NRS Score) | Baseline, Week 2, Week 4, and Week 8
  Change in Numeric Rating Scale (NRS) for pain intensity from baseline to week 8 following the MOVE (Movement-Oriented Velocity of Engagement) rehabilitation program. Participants rated pain on a 0-10 scale where 0 = no pain and 10 = worst possible pain.

SECONDARY OUTCOMES:
Functional Improvement (LEFS / UEFI Score) | Baseline, Week 2, Week 4, Week 8
  Change in Lower Extremity Functional Scale (LEFS) or Upper Extremity Functional Index (UEFI) from baseline to week 8, reflecting mobility and activity performance improvement post-MOVE intervention.
Balance and Postural Stability (Timed Single-Leg Stance Test) | Baseline, Week 4, Week 8
  Improvement in single-leg stance duration and balance control across sessions as measured by standardized postural tests.
Participant Perceived Recovery (Global Rating of Change Scale) | Week 8
  Participants rate overall improvement on a 7-point Global Rating of Change (GROC) scale at week 8 to capture subjective recovery perception.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - BodyGNTX Fitness Institute, Columbus, Ohio
  - MMSx AUTHORITY (COORDINATING CENTER), Powell, Ohio
- India (2):
  - Indian Institute of Kinesiology & Biomechanics Science (IIKBS), Burhānpur, Madhya Pradesh
  - GFFI Fitness Academy, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: No
De-identified participant data are stored securely at MMSx Authority Clinical Research Division and affiliated academic centers (BodyGNTX USA, GFFI India, IIKBS). Data will not be shared publicly but may be used in aggregate form for institutional publications.

DOCUMENTS (2):
  • Study Protocol (2024-06-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT07220200/Prot_000.pdf
  • Informed Consent Form (2024-06-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT07220200/ICF_001.pdf